CLINICAL TRIAL: NCT02985684
Title: GORE® CARDIOFORM ASD Occluder Clinical Study: A Study to Evaluate Safety and Efficacy in the Treatment of Transcatheter Closure of Ostium Secundum Atrial Septal Defects (ASDs) - The Gore ASSURED Clinical Study
Brief Title: Safety and Efficacy Study of Transcatheter Closure of Ostium Secundum ASDs
Acronym: ASSURED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASD 15-04
Record Dates: First submitted 2016-11-28; First posted 2016-12-07 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Atrial Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device (Experimental): ASD closure with the GORE® CARDIOFORM ASD Occluder
  Interventions: Device: GORE® CARDIOFORM ASD Occluder

INTERVENTIONS:
Device: GORE® CARDIOFORM ASD Occluder — Percutaneous Atrial Septal Defect Closure

SUMMARY:
Evaluate the safety and efficacy of the GORE® CARDIOFORM ASD Occluder in the percutaneous closure of ostium secundum atrial septal defects (ASDs)

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm clinical study comparing outcomes with the GORE® CARDIOFORM ASD Occluder to performance goals derived from clinical investigation outcomes for devices indicated for ASD closure.

ELIGIBILITY:
Inclusion Criteria:

All responses must be Yes to be eligible:

1. Patient has an ostium secundum ASD with evidence of left-to-right shunt and right ventricular volume overload.
2. Patient has a defect size 8-35 mm as measured directly by stop-flow balloon sizing.
3. Patient vasculature can accommodate the delivery system and procedural accessories.
4. Patient can accommodate TEE or intracardiac echocardiography (ICE) probe for implant procedure.
5. Patient is judged by the implanting physician to have adequate septal rims to retain the study device.
6. Patient (or legal guardian, if patient is a minor) will voluntarily sign a Patient Informed Consent Form (ICF) specific to the study. The Patient ICF must be reviewed and approved in a manner that complies with requirements of the hospital's Institutional Review Board (IRB).
7. Patient (and legal guardian, if patient is a minor) is physically and mentally willing to comply with all study follow-up requirements through 36 months, including routinely scheduled diagnostic testing and physical examinations.

Exclusion Criteria:

All responses must be No to be eligible:

1. Patient has significant known pre-existing electrophysiologic or structural cardiovascular defect, or other comorbidities that could elevate morbidity or mortality beyond what is common for ASD or would require surgical treatment within three (3) years of device placement. Examples include, but are not limited to, large ventricular septal defect, hypoplastic left heart syndrome, coarctation, univentricular heart or tricuspid atresia, pulmonary hypertension, coronary artery disease, valvular or myocardial dysfunction, and other congenital heart disease requiring surgical repair.
2. Patient has systemic or inherited conditions that would significantly increase risk of major morbidity and mortality during the term of the study. Examples include endocarditis, cancer, degenerative neuromuscular disorder, cardiomyopathy, and any condition expected to result in significant deterioration of health within three (3) years of the index procedure.
3. Patient has anatomy where the size or position of the occluder would interfere with other intracardiac or intravasculature structures, such as cardiac valves or pulmonary veins.
4. Patient has active endocarditis, other infections producing bacteremia, or has known sepsis within one month of planned implantation, or any other infection that cannot be treated successfully prior to device placement.
5. Patient has known intracardiac thrombi.
6. Patient has an uncontrolled arrhythmia with evidence of arrhythmia control failure within the past 90 days (e.g., supraventricular tachycardia while under rate control or atrial fibrillation while under rhythm control) or requires electrophysiology study or concomitant intervention with device placement.
7. Patient is awaiting a procedure that requires trans-septal left atrial access within 6 months of implant procedure.
8. Patient has a history of stroke resulting in a significant morbidity or disability.
9. Patient is pregnant or lactating at time of screening.
10. Patient has contraindication to antiplatelet and anticoagulant medications.
11. Patient has elevated pulmonary vascular resistance (PVR) which in the opinion of the implanting physician precludes safe defect closure.
12. Patient has multiple defects based on screening imaging and stop-flow balloon sizing that would require placement of more than one device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sommer, MD, Principal Investigator — Columbia University of New York; Matthew Gillespie, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (22):
- United States (22):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California-Los Angeles, Los Angeles, California
  - The Children's Hospital of Colorado, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Nicklaus Children's Hospital, Miami, Florida
  - Children's Healthcare at Egleston, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Hospital & Regional Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qureshi AM, Sommer RJ, Morgan G, Paolillo JA, Gray RG, Love B, Goldstein BH, Sugeng L, Gillespie MJ; GORE ASSURED Clinical Trial Investigators. Long-Term Results of the Atrial Septal Defect Occluder ASSURED Trial for Combined Pivotal/Continued Access Cohorts. JACC Cardiovasc Interv. 2024 Oct 14;17(19):2274-2283. doi: 10.1016/j.jcin.2024.07.013. Epub 2024 Sep 18. PMID 39297855

RESULTS

PARTICIPANT FLOW:
Period: 6-Month Clinical Success Evaluation
Arm/Group | Device
Started | 125
Completed | 120
Not Completed | 5
Not completed — Missed Echocardiograph | 5
Period: 6-Month Closure Success Evaluation
Arm/Group | Device
Started | 120
Completed | 112
Not Completed | 8
Not completed — Technical Failure (No Device) | 5
Not completed — Device Removal | 3

BASELINE CHARACTERISTICS:
Population: All enrolled pivotal subjects
Arm/Group | Device
Number analyzed (Participants) | 125
Age, Continuous [Median (Full Range); unit: years] | 12.3 [2.9 to 84.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 6
  White | 83
  More than one race | 0
  Unknown or Not Reported | 28
Region of Enrollment [Number; unit: participants]
  United States | 125
Height [Median (Full Range); unit: cm] | 148 [85 to 191]
Weight [Median (Full Range); unit: kg] | 41.5 [12.0 to 105.2]
Hypercholesterolemia [Count of Participants; unit: Participants]
  Current | 8
  Previous/Never | 117
Hypertension [Count of Participants; unit: Participants]
  Current | 6
  Previous/Never | 119
Diabetes Mellitus [Count of Participants; unit: Participants]
  Current | 2
  Previous/Never | 123
Nicotene Use [Count of Participants; unit: Participants]
  Within past year | 1
  >1 year ago | 2
  Never | 122
Headaches or Migraines [Count of Participants; unit: Participants]
  Current | 7
  Previous | 9
  Never | 109
Cardiac Arrhythmia History [Count of Participants; unit: Participants] | 17
Stop Flow Balloon Defect Size [Median (Full Range); unit: mm] | 17 [8 to 30]
Multiple Fenestrations [Count of Participants; unit: Participants] | 18
Atrial Septal Aneurysm [Count of Participants; unit: Participants] | 6
Septal Length [Median (Full Range); unit: mm] | 39 [21 to 65]
Anterior-Superior Aortic Rim Length [Median (Full Range); unit: mm] | 4 [0 to 27]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With 6-Month Closure Success
Description: Among subjects with technical success, the number of subjects with clinical residual defect status of occluded or clinically insignificant as determined by the Echo Core Lab at the 6-month evaluation.
Time Frame: 6 months
Population: Pivotal subjects with technical success and 6-month clinical residual defect status evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 112
Participants | 112
Statistical Analysis 1: Comparison: Device; Test null hypothesis of equal or lesser proportion with 6-month closure success compared to a performance goal (PG). H0: P ≤ 0.88 vs H1: P > 0.88, where P is the true proportion of subjects with 6-month closure success and 0.88 is the PG derived from clinical study outcomes for devices indicated for ASD closure. N=103 subjects provide ≥95% power to exclude PG with 95% confidence if P=0.98 under H1; Test type: Other — Acceptable performance: favorably exclude PG=0.88 with 95% confidence. Expected 6-month closure success proportion = 0.98. Acceptable performance margin = 0.10. PG = 0.98 - 0.10 = 0.88; p < 0.0001, Binomial test (exact) — A priori 1-sided alpha = 0.05. If test rejects H0, then test primary outcome 2 (clinical success) at 1-sided alpha = 0.05; otherwise testing stops with failure to reject both primary outcome null hypotheses; Binomial proportion = 1.0, 95% CI 1-sided [lower limit 0.974] — Exact 1-sided confidence interval lower bound from Clopper-Pearson method

2. Primary Outcome: Number of Subjects With 6-Month Composite Clinical Success
Description: Among subjects with attempted study device closure, the number of subjects who satisfy all of the following components:
  1. Technical Success: Successful deployment and retention at conclusion of index procedure of a GORE® CARDIOFORM ASD Occluder
  2. Safety Success:
     * Freedom from any Serious Adverse Event (SAE) related to the device or procedure as adjudicated by the Independent Data Review Board (IDRB) through 30 days post-procedure
     * Freedom from device events (post-procedure embolization, device removal, or other device reintervention) from completion of the implant procedure through 6 months (180 days) post-procedure
  3. Closure Success: A clinical residual defect status of occluded or clinically insignificant as determined by the Echo Core Lab at the 6-month evaluation
Time Frame: 6 months
Population: All enrolled pivotal subjects with 6-month clinical success evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 120
Participants | 108
Statistical Analysis 1: Comparison: Device; Test null hypothesis of equal or lesser proportion with 6-month clinical success compared to a performance goal (PG). H0: P ≤ 0.76 vs H1: P > 0.76, where P is the true proportion of subjects with 6-month clinical success and 0.76 is the PG derived from clinical study outcomes for devices indicated for ASD closure. N=112 subjects provide 95% power to exclude PG with 95% confidence if P=0.88 under H1; Test type: Other — Acceptable performance: favorably exclude PG=0.76 with 95% confidence. Expected 6-month clinical success proportion = 0.88. Acceptable performance margin = 0.12. PG = 0.88 - 0.12 = 0.76; p < 0.0001, Binomial test (exact) — A priori 1-sided alpha = 0.05. If test of primary outcome 1 rejects H0, then test at 1-sided alpha = 0.05; otherwise no testing of this primary outcome and failure to reject null hypothesis; Binomial proportion = 0.90, 95% CI 1-sided [lower limit 0.843] — Exact 1-sided confidence interval lower bound from Clopper-Pearson method

3. Secondary Outcome: Number of Subjects With Technical Success
Description: Among subjects with attempted study device closure, the number of subjects with successful deployment and retention at conclusion of index procedure of a GORE® CARDIOFORM ASD Occluder
Time Frame: During procedure; median duration 67 minutes
Population: All pivotal subjects enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 125
Participants | 120

4. Secondary Outcome: Number of Subjects With Procedure Success
Description: Among subjects with attempted study device closure, the number of subjects with technical success and measured residual defect status of occluded, small, or moderate of the target ASD at conclusion of index procedure
Time Frame: During procedure; median duration 67 minutes
Population: All pivotal subjects enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 125
Participants | 120

5. Secondary Outcome: Number of Subjects With 30-day IDRB-adjudicated Device- or Procedure-related SAE
Description: Among subjects with attempted study device closure, the number of subjects experiencing one or more device- or procedure-related serious adverse events (SAEs) within 30 days post-index procedure as adjudicated by the Independent Data Review Board (IDRB)
Time Frame: 30 days
Population: All enrolled pivotal subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 125
Participants | 6

6. Secondary Outcome: Measured Residual Target Defect Size
Description: Measured residual defect size (in millimeters) as determined by the Echo Core Lab at the 6-month evaluation.
Time Frame: 6 months
Population: Pivotal subjects with technical success and 6-month measured residual defect status evaluation
Measure: Median (Full Range); unit: mm
Arm/Group | Device
Number analyzed (Participants) | 112
mm | 0.0 [0.0 to 4.6]

7. Secondary Outcome: Number of Subjects With Clinically Significant New Arrhythmia
Description: The number of subjects with any new arrhythmia (documented on ECG) requiring hospitalization, initiation of new long-term medical therapy (persisting > 45 days), or any post-index procedure cardioversion or intervention (pacemaker, ablation, etc.) in subjects without prior history of arrhythmia, as adjudicated by the Independent Data Review Board
Time Frame: 6 months
Population: All pivotal subjects enrolled -- prior history of arrhythmia reported on the medical history form does not preclude assessment for, and finding of, clinically significant new arrhythmia from adjudication by the Independent Data Review Board
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 125
Participants | 6

8. Secondary Outcome: Number of Subjects With Wire Frame Fracture
Description: Among subjects with technical success, the number of subjects with wire frame fracture as determined by fluoroscopy at the 6-month evaluation.
Time Frame: 6 months
Population: Pivotal subjects with technical success and 6-month fluoroscopy evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 104
Participants | 37

ADVERSE EVENTS:
Time Frame: 6 months (180 days)
Arm/Group | Device
All-Cause Mortality (participants affected / at risk) | 0/125
Serious Adverse Events (participants affected / at risk) | 8/125
Other Adverse Events (participants affected / at risk) | 57/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=125)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Device embolisation (General disorders) | 2 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1)
Thrombosis in device (Product Issues) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=125)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (5)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Enlarged uvula (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Catheter site haematoma (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 6 (6)
Pyrexia (General disorders) | 2 (2)
Jaundice (Hepatobiliary disorders) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Trichomoniasis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Vaginal infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1)
Heart rate decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 6 (7)
Migraine (Nervous system disorders) | 1 (3)
Seizure (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal exudate (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT02985684/Prot_003.pdf
  • Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT02985684/SAP_001.pdf